CLINICAL TRIAL: NCT06683690
Title: TGF β 1 Expression Related Gene Polymorphism and Their Association With Clinical Types of Leprosy
Brief Title: TGF β 1 Expression Related Gene Polymorphism
Status: Recruiting | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Gehad Adel Abd El-Sabour Mohammed, Specialist of Dermatology, Aswan University
Other Study IDs: Gehad Adel Abd El-Sabour
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-07

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Leprosy Patients: About 30 patients affected with Leorosy
  Interventions: Procedure: Measurement of TGF- β1 in leprosy patients
- Group B: Healthy People: About 30 Healthy participants
  Interventions: Procedure: Measurement of TGF- β1 in leprosy patients

INTERVENTIONS:
Procedure: Measurement of TGF- β1 in leprosy patients — Study TGF- β1gene polymorphism in leprosy patients, and Correlate their results with different types of leprosy before and after treatment.

SUMMARY:
Leprosy is one of the oldest human infectious diseases. It is a chronic infectious contagious, granulomatous disease caused by intracellular bacillus.

Mycobacterium leprae, this chronic granulomatous disease presents symptoms that mainly affected the skin, the nervous system and the reticuloendothelial system, also other systems can be affected, such as the upper respiratory tract, bones and joints, eyes and adrenal glands.

TGF- β is a pleiotropic cytokine that employs several functions on different types of cells. The effect of other cytokines may finally modulate the cellular response in the presence of TGF- β, causing a different effect depending on the activation state of the cell involved. In addition, TGF- β promotes the healing of inflamed tissue through the stimulation and regulation of extracellular matrix by fibroblasts, in addition to inducing the proliferation of endothelial cells required for angiogenesis. Thus, TGF- β is able to regulate the expression of other growth factors, increasing their level of activity.

DETAILED DESCRIPTION:
The spectrum of clinical and histopathological manifestations reflects the immune response elicited by the microorganism in the host leprosy classified into polar groups:

Lepromatous (LL) and Tuberculoid (TT); and borderline spectrum: Borderline Tuberculoid (BT), Borderline Borderline (BB) and Borderline Lepromatous (BL). This classification, proposed by Ridley and Jopling This classification widely used in clinical, immunological, microbiological, and histopathological aspects. While The World Health Organization classifies leprosy clinically as multibacillary and paucibacillary, according to the number of skin lesions and nerve involvement.

In the tuberculoid form of leprosy (paucibacillary), the individual manifests an intense cell-mediated immune response that prevents proliferation of the bacillus, whereas the cell-mediated immune response is compromised in the lepromatous form (multibacillary) contributing to multiplication of the bacillus. In the intermediate forms,the patients exhibit characteristics that vary between the two types.

Leprosy is measured the first disease to be categorized based on the host's immune response. The clinical symptoms of leprosy vary from one patient to another based on the spectrum of disease but more importantly on the type of host's immune response to the bacteria. Both innate and acquired immune responses have been associated with leprosy, but the disease is typically described by the side of a Th1/Th2 response.

Patients with TT are decided by a relevant T-cell immune response, including interleukin-2 (IL-2), IL-4, IL-6, IL-10, interferon-γ (IFN-γ), tumor necrosis factor (TNF), and IL-17 and lymphotoxin, marked by some neural or cutaneous lesions with a few or no bacilli.

Infected macrophages are activated by IFN- γ and clonal expansion of T cells is induced by IL-2 which, in turn, leads to an increase in IFN- γ production. Tumor necrosis factor alpha (TNF- α) also plays a role in the Th1 response. This cytokine contributes to the maintenance of this pattern and acts in synchronism with IFN- γ in the activation of infected macrphages, developing a significant mechanism for the maintenance of the cell-mediated immune response.

In contrast, patients with LL show a superior humoral immune response, characterized by multiple lesions, elevated bacterial load, and reduced lymphocyte production develop a Th2 immune response characterized by intense production of transforming growth factor beta (TGF- β), IL-4, IL-5 and IL-10.

These cytokines induce an incompetent immune response characterized by the high production of antibodies that apply no protective effect against the bacterium.

IL-4 exerts an immunosuppressive effect that leads to an increase in bacterial proliferation and inhibits the proliferation of T cells and monocytes, the expression of CD14 on monocytes and the production of TNF- α, in addition to blocking the synthesis of nitric oxide which is essential for the destruction of intracellular microorganisms. In the 21st century, studies using modern genetic methods such as candidate gene association studies (CGASs) and genome wide association studies (GWASs) have gradually confirmed that the host genetic background play important role in the development of leprosy, and many leprosyassociated variants or genes have been reported. Most leprosy-associated genes are immune related, which is consistent with the finding that leprosy is caused by infection with pathogen.

TGF β1 plays roles in the suppression of T cell responses, inhibiting both IFN γ and IL-2 expression, and has the ability to inhibit the lytic activity of macrophages by suppressing the production of intermediate oxygen-reactive and nitrogen-reactive factors, leading to the progression of infection. So, the production of TGF β1 by macrophages in LL and BL skin lesions, probably as part of the M. leprae evasion mechanism.

Experimental studies on these pathogenic agents have demonstrated a role of TGF- β1 as a suppressor of macrophages. TGF-β1 production in lepromatous patients, which contributes to the anti-inflammatory situation and bacillary persistence observed

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with leprosy.
* Age above 18 years.
* patients on multidrug therapy of leprosy.

Exclusion Criteria:

* Patients with other dermatological disease.
* Patients with leprosy reaction.
* Pregnancy and lactation.
* Patients with autoimmune disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include (30) leprosy patients and (30) normal control , selected from the outpatient clinic of the Dermatology, Venereology, and Andrology Department, at Aswan University Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Detection of serum TGF β1 | One Year
  Detection of serum TGF β1 in leprosy patients and Correlate them with different clinical types of leprosy by taking Blood Samples will be collected from the patients to detect TGF β1gene by DNA extraction and SNP genotyping - Genomic DNA will be extracted from peripheral blood samples, then the polymorphism of the TGF β1 gene marker will be selected, The Blood Samples will be collected from the patients before and after treatment with multidrug therapy of leprosy to detect the level of TGF β1 concentrations by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam Ali El Taieb, Professor, Study Chair — Dermatology, Venereology and Andrology. Faculty of Medicine, Aswan University; Abdallah Mahmoud Abdallah, Professor, Study Director — Biochemistry and Molecular Biology. Faculty of Medicine, Aswan University
Locations (1):
- Aswan Universit Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided